CLINICAL TRIAL: NCT04916613
Title: A Double-blind Randomised Phase III Trial Evaluating the Efficacy of ADT +/- Darolutamide in de Novo Metastatic Prostate Cancer Patients With Vulnerable Functional Ability and Not Elected for Docetaxel or Androgen Receptor Targeted Agents
Brief Title: ADT +/- Darolutamide in de Novo Metastatic Prostate Cancer Patients With Vulnerable Functional Ability (PEACE6-Vulnerable)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UC-GTG-2006; 2020-003663-26 (EudraCT Number)
Record Dates: First submitted 2021-06-04; First posted 2021-06-07 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — darolutamide; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Phase III, international, multicenter, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded placebo controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADT + darolutamide (Experimental): ADT + darolutamide 600 mg po bid
  Interventions: Drug: Darolutamide 300 mg; Drug: Androgen deprivation therapy
- ADT + placebo (Placebo Comparator): ADT + placebo po bid
  Interventions: Drug: Placebo; Drug: Androgen deprivation therapy

INTERVENTIONS:
Drug: Darolutamide 300 mg — 600 mg po, b.i.d.
  Other Names: Nubeqa®
  Arms: ADT + darolutamide
Drug: Placebo — po, b.i.d.
  Arms: ADT + placebo
Drug: Androgen deprivation therapy — Use according to local standard of care
  Other Names: ADT

SUMMARY:
This is a Phase III, international, multicentre, randomised, double-blinded placebo controlled trial, evaluating the efficacy and safety of ADT +/- darolutamide in castration-naïve de novo metastatic prostate cancer patients with vulnerable functional ability who have not elected for docetaxel or other androgen receptor pathway inhibitors.

DETAILED DESCRIPTION:
This is a Phase III, international, multicentre, randomised, double-blinded placebo controlled trial, evaluating the efficacy and safety of ADT +/- darolutamide in castration-naïve de novo metastatic prostate cancer patients with vulnerable functional ability who have not elected for docetaxel or other androgen receptor pathway inhibitors. The study plans to enroll 300 patients who will be randomized (1:1) to receive either: (i) Experimental arm: ADT + darolutamide 600 mg po bid, or (ii) Control arm: ADT + placebo po bid. Response to treatment will be assessed according to the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria (Scher, 2016). Treatment will be continued until radiographic disease progression. Treatment may also be terminated at the initiative of either the patient or the investigator for any reason that would be beneficial to the patient, including: unacceptable toxicity, intercurrent conditions that preclude continuation of treatment, or patient request. Following treatment discontinuation patients will enter the follow-up period and will be monitored for up to 10 years with regards to survival status, subsequent antineoplastic treatments and the status of ongoing adverse events (AEs) and/or new investigational product related AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form prior to any trial specific procedures.
2. Men with histologically or cytologically confirmed adenocarcinoma of the prostate.
3. Aged ≥18 years old at the time of signing informed consent.
4. De novo metastatic disease defined by clinical or radiological evidence of metastases.

   Note: For patients with nodal metastases only, only patients with extra-pelvic enlarged lymph nodes (lymph nodes located above the iliac bifurcation) can be included if they have either:
   * At least one extra-pelvic lymph node ≥2 cm
   * At least one extra-pelvic lymph node ≥1 cm if the patients also have at least one pelvic lymph node ≥2 cm
5. Measurable disease or bone lesions that are evaluable according to PCWG3 criteria.
6. Ineligible for treatment with all of the following drugs: docetaxel, abiraterone, enzalutamide, apalutamide; AND meets at least one of the following frailty criteria:

   1. Activities of daily living (ADL) assessment (excluding urinary incontinence question) score 3 or 4/5, or;
   2. 4-Instrumental activities of daily living (4-IADL) assessment score 2 or 3/4, or;
   3. A Grade 3 event on the Cumulative Illness Score Rating-Geriatrics (CISR-G) questionnaire, or;
   4. Body mass index (BMI) ≤21 kg/m² and/or >5% weight loss in the last 6 months, or;
   5. Timed up and go test (TUG) >14 sec. Nota Bene: Regarding CISR-G assessment, more specifically genitourinary scoring, score N°4 is not applicable.
7. Adequate bone marrow function: haemoglobin ≥80 g/L, white blood cells ≥3.0 x10⁹/L and platelets ≥80 x10⁹/L.
8. Adequate liver function: alanine aminotransferase (ALT) <2 x upper limit of normal (ULN) and bilirubin <1.5 x ULN, (or if bilirubin is between 1.5-2 x ULN, they must have a normal conjugated bilirubin). For patients with documented liver metastasis, ALT <5 x ULN is acceptable.
9. Adequate renal function: calculated creatinine clearance >30 ml/min (using the Modification of Diet in Renal Disease [MDRD] or Chronic Kidney Disease Epidemiology Collaboration [CKD EPI) method).
10. For sexually active men, agreement to use adequate contraception for the duration of trial participation and up to 2 weeks after completing study treatment.
11. Affiliated to the social security system or in possession of equivalent private health insurance (according to local regulations for participation in clinical trials).
12. Willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

1. Three or more Grade 3, or any Grade 4 events on the CISR-G questionnaire. Nota Bene: (Regarding CISR-G assessment, more specifically genitourinary scoring, score N°4 is not applicable).
2. Eastern Cooperative Oncology Group (ECOG) performance status score ≥3.
3. Hypertension not controlled by an anti-hypertensive treatment (systolic blood pressure [BP] ≥160 mmHg or diastolic BP ≥95 mmHg; 3 consecutive measures taken 5 minutes apart).
4. Acute toxicities of prior treatments and procedures not resolved to grade ≤1 or baseline before randomisation, with the exception of hot flushes and erectile dysfunction.
5. Previous systemic treatment for prostate cancer, except less than 12 weeks of ADT and/or an old-generation AR inhibitor.
6. Severe or uncontrolled concurrent disease, infection or co-morbidity.
7. Known hypersensitivity to the study treatment or any of its ingredients.
8. Major surgery within 28 days before randomisation.
9. Any of the following within 6 months before randomisation: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft; congestive heart failure New York Heart Association (NYHA) Class III or IV.
10. Prior malignancy ≤3 years before study enrolment. Adequately treated basal cell or squamous cell carcinoma of skin or superficial bladder cancer that has not spread behind the connective tissue layer (i.e., pTis, pTa, and pT1) is allowed, as well as any localized cancer for which treatment has been completed ≥6 months before randomisation and from which the subject has been disease-free, or for which the risk of relapse is less than 30%, as well as early stage chronic lymphocytic leukaemia that does not require any specific treatment.
11. Inability to swallow oral medications.
12. Gastrointestinal disorder or procedure that can be expected to interfere significantly with the absorption of study treatment.
13. Known to have active viral hepatitis, active human immunodeficiency virus (HIV) or chronic liver disease at screening.
14. Treatment with any investigational product within 28 days before randomisation.
15. Concurrent participation in another clinical trial involving an investigational product (patients enrolled in non-experimental trials with no modification of the standard of care can be included).
16. Individual deprived of liberty or placed under the authority of a tutor.
17. Significantly altered mental status prohibiting the understanding of the study or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule or any condition that, in the opinion of the investigator, would preclude participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2037-09 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression-free survival | From randomisation to radiographic progression or death, up to 18 months
  Time from randomisation to radiographic progression according to the Prostate Cancer Working Group 3 (PCWG3) criteria or death, whichever occurs first

SECONDARY OUTCOMES:
Castration-resistant prostate cancer-free survival | From randomisation to onset of CRPC or death, up to 18 months
  Time from randomisation to onset of castrate resistant prostate cancer (CRPC) according to PCWG3 criteria, or death, whichever occurs first
Clinical progression-free survival | From randomisation to clinical progression or death, up to 18 months
  Time from randomisation to first occurrence of any one of the following:
  (i) Cancer pain deterioration (2-point deterioration from baseline according to the Brief Pain Inventory - Short Form [BPI-SF] questionnaire; initiation of opioid therapy, or a ≥30% increase in opiate use) (ii) Any deterioration of physical function measured using the 4-IADL assessment tools (Lawton, 1969) (iii) A deterioration in ECOG performance status of at least 2 points from baseline (iv) Death from any cause.
Overall survival | From randomization to death from any cause, up to 10 years.
  Time from randomisation to the time of death from any cause
Frequency and severity of adverse events | From inclusion until 100 days after last dose of investigational product
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders
Time to worsening in prostate cancer-related urinary symptoms | On treatment day 1 and every 120 days during first years of treatment and every 180 days thereafter if treatment is continued for more than 1 year
  Time from randomisation to first increase from baseline of greater or equal to 8 points in the urinary symptom scale/score (PRURI) measured using the prostate cancer module of the EORTC quality of life questionnaire (EORTC-QLQ-PR25).
  This EORTC prostate cancer specific questionnaire is intended to supplement the QLQ-C30. The prostate cancer module is a 25-item questionnaire designed for use among patients with localized and metastatic prostate cancer. It includes subscales assessing urinary symptoms (9 items), bowel symptoms (4 items), treatment-related symptoms (6 items) and sexual functioning (6 items). Using a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), patients indicate the degree to which they have experienced symptoms.
Time to next symptomatic skeletal event | From randomisation to occurence of a skeletal event, up to 18 months
  Time from randomisation until first occurrence of one of the following: a symptomatic fracture, radiation or surgery to bone or a spinal cord compression
Complete prostate specific antigen (PSA) response | At 6 months
  Defined according to PCWG3 criteria as PSA ≤ 0.2 ng/ml
Prostate cancer-specific survival | From randomization to death from prostate cancer, up to 10 years.
  Time from randomisation to the date of death due to prostate cancer (deaths due to other causes will be censored)
Time to first subsequent systemic anti-cancer therapy (SACT) | From randomization up to 10 years.
  Time from randomisation to the date of initiation of any SACT for CRPC, following initiation of the study treatment
Second line radiographic progression-free survival | From randomization up to 10 years.
  Time from the date of initiation of a second SACT for CRPC to radiographic progression or death, whichever occurs first.
Second line overall survival | From randomization up to 10 years.
  Time from the date of initiation of a second SACT for CRPC to death
Progression-free survival after next line of treatment (PFS2) | From randomization up to 10 years.
  Time from randomisation to second objective disease progression, or death from any cause, whichever first
Geriatric status | At baseline and every 120 days during first years of treatment and every 180 days thereafter if treatment is continued for more than 1 year
  Evaluated using the G-CODE (Paillaud, 2018), a core set of commonly used tools/items for geriatric assessment which has been validated for the collection of geriatric data in clinical cancer trials of older adults, enabling comparison across trials. The tools/items proposed in G-CODE are:
  (i) Social assessment: living alone or support requested to stay at home; (ii) Functional autonomy: Activities of Daily Living (ADL) questionnaire and short instrumental ADL questionnaire (4-IADL); (iii) Mobility: Timed Up and Go test; (iv) Nutrition: weight loss during the past 6 months and body mass index; (v) Cognition: Mini-Cog test; (vi) Mood: mini-Geriatric Depression Scale; (vii) Comorbidity: updated Charlson Comorbidity Index.
Time to deterioration for EORTC QLQ-PR25 symptom subscales | On treatment day 1 and every 120 days during first years of treatment and every 180 days thereafter if treatment is continued for more than 1 year
  Defined as the first decline in the HRQoL score from baseline equal to or greater than the minimally important difference (MID; a measure of clinical significance) defined as half the standard deviation of the baseline value for each subscale. The prostate cancer module QLQ-PR25 is a 25-item questionnaire designed for use among patients with localized and metastatic prostate cancer. It includes subscales assessing urinary symptoms (9 items), bowel symptoms (4 items), treatment-related symptoms (6 items) and sexual functioning (6 items). Using a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), patients indicate the degree to which they have experienced symptoms.
Health related quality of life questionnaire EORTC-QLQ-C30 | On treatment day 1 and every 120 days during first years of treatment and every 180 days thereafter if treatment is continued for more than 1 year
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Health related quality of life questionnaire EORTC-QLQ-PR25 | On treatment day 1 and every 120 days during first years of treatment and every 180 days thereafter if treatment is continued for more than 1 year
  This EORTC prostate cancer specific questionnaire is intended to supplement the QLQ-C30.
  The prostate cancer module is a 25-item questionnaire designed for use among patients with localized and metastatic prostate cancer. It includes subscales assessing urinary symptoms (9 items), bowel symptoms (4 items), treatment-related symptoms (6 items) and sexual functioning (6 items). Using a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), patients indicate the degree to which they have experienced symptoms.
Health related quality of life questionnaire Brief Pain Inventory - Short Form (BPI-SF) | On treatment day 1 and every 120 days during first years of treatment and every 180 days thereafter if treatment is continued for more than 1 year
  The Brief Pain Inventory is a self reporting tool to assess the severity of pain and the impact of pain on daily functions in patients with chronically painful diseases or conditions such as cancer, osteoarthritis and low back pain, or with pain from acute conditions such as postoperative pain. The Short Form of the questionnaire (BPI-SF) has been specifically developed for clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Baciarello, MD, Principal Investigator — San Camillo-Forlanino hospital, Italy; Karim Fizazi, MD, Principal Investigator — Gustave Roussy Cancer Campus, France
Locations (90):
- Belgium (4):
  - Grand Hopital de Charleroi - site Notre Dame, Charleroi
  - Groupe Jolimont - Hôpital De Jolimont, Haine-Saint-Paul
  - CHU UCL NAMUR - Site STE. ELISABETH, Namur
  - Clinique Saint Pierre, Ottignies
- France (46):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Cote basque, Bayonne
  - CHU Besançon - Hopital Jean Mijoz, Besançon
  - Centre Institut Bergonié, Bordeaux
  - Clinique Pasteur, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier Métropole Savoie, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - APHP - Hôpital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHU de la Martinique - Hôpital Albert Clarac, Fort-de-France
  - CHU Grenoble, Grenoble
  - Centre CHV Vendée, La Roche-sur-Yon
  - CHU le MANS, Le Mans
  - Centre Oscar Lambret, Lille
  - Polyclinique de Limoges, Limoges
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Antoine Lacassagne, Nice
  - CHU Nîmes, Nîmes
  - Centre Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Hospices Civils de Lyon -Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Pôle Régional de Cancérologie, Poitiers
  - CH Annecy Genevois, Pringy
  - CHIC Quimper, Quimper
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier Rodez, Rodez
  - CHU Saint-Etienne, Saint-Etienne
  - Hôpital Privé de la Loire, Saint-Etienne
  - CHP Centre Saint Grégoire, Saint-Grégoire
  - Hôpital Instruction des Armées - BEGIN, Saint-Mandé
  - Clinique Sainte Anne - Strasbourg Oncologie Libérale, Strasbourg
  - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Hôpital FOCH, Suresnes
  - Centre Hospitalier Intercommunal de Toulon-La Seyne - Hôpital Ste Musse, Toulon
  - IUCT Oncopole, Toulouse
  - Clinique Pasteur ONCORAD, Toulouse
  - CHRU de Tours -Hôpital Bretonneau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy Center, Villejuif
- Germany (3):
  - Universitätsmedizin Essen Hufelandstraße, Essen
  - University cancer center Hamburg-Eppendorf Martinistraße, Hamburg
  - Universitätsklinikum Münster Klinik für Urologie und Kinderurologie Albert-Schweitzer-Campus 1 Gebäude A1, Münster
- Ireland (4):
  - St Vincent's University Hospital, Dublin
  - Tallaght university Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
- Italy (10):
  - University of Bari, Policlinico, Bari
  - FPO IRCCS Candiolo Turin, Candiolo
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola
  - Fondazione IRCSS Istituto Nazionale Tumori, Milan
  - istituto tumori Fondazione "G.Pascale", Napoli
  - Azienda Ospedaliera S. Camillo-Forlanini, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas - IRCCS, Rozzano
  - UOC Oncologia Medica, Syracuse
  - Santa Chiara Hospital, Trento
- Netherlands (2):
  - Albert Schweizer Hospital, Dordrecht
  - Radboudumc - Dutch Uro-Oncology Study Group (DUOS), Nijmegen
- Romania (4):
  - Institutul Oncologic Prof Dr Al Trestioreanu Bucuresti, Bucharest
  - Amethyst Radiotherapy Center Cluj SRL, Cluj-Napoca
  - Institul Oncologic Cluj-Napoca, Cluj-Napoca
  - OncoHelp Hospital, Timișoara
- Narodny Onkologicky Institut, Bratislava, Slovakia
- Spain (9):
  - Institut Catala d'Oncologia, Badalona-Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology. Vall d'Hebron University Hospital, Barcelona
  - Institut Català d'Oncologia de Girona, Girona
  - Centro Integral Oncologico HM Clara Campal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Althaia, Xara Assistencial Universitaria Mansera, Manresa
  - Fundacion Instituto Valenciano De Oncologia, Valencia
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Malmo
- Switzerland (5):
  - Istituto Oncologico della Svizzera Italiana (IOSI) - Ospedale S.Giovanni, Bellinzona
  - Kantonsspital Graubünden, Onkologie/ Hämatologie, Chur
  - Cantonal Hospital St.Gallen, Sankt Gallen
  - Istituto Oncologico della Svizzera Italiana (IOSI) - Ospedale Italiano di Lugano, Viganello
  - Universitätsspital Zürich - Onkologie, Zurich

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon request to the sponsor
Supporting Information: Study Protocol, CSR
Time Frame: After primary analysis until end of trial
Access Criteria: Steering committee approval